CLINICAL TRIAL: NCT03073967
Title: A Randomized, Open Label, Multi-center, Comparative Trial, to Assess the Efficacy and Safety of Pritelivir for the Treatment of Acyclovir-resistant Mucocutaneous HSV (Herpes Simplex Virus) Infections in Immunocompromised Subjects (PRIOH-1)
Brief Title: Trial on Efficacy and Safety of Pritelivir Tablets for Treatment of Acyclovir-resistant Mucocutaneous HSV (Herpes Simplex Virus) Infections in Immunocompromised Subjects
Acronym: PRIOH-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AiCuris Anti-infective Cures AG (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIC316-03-II-01
Expanded Access: NCT05844436 (Available)
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: HSV Infection
MeSH Terms: conditions — Herpes Simplex | interventions — pritelivir; Foscarnet; Cidofovir; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part C, Pritelivir (Experimental): Oral tablets, 100mg/day (400mg loading dose on day 1) for up to 28 days and potential prolongation for up to additional 14 days
  Interventions: Drug: Pritelivir
- Part C, (Active Comparator): Investigator's Choice:
  Foscarnet iv, 40 mg/kg tid or 60mg/kg bid or Cidofovir iv, 5 mg/kg body weight given once weekly or Cidofovir 1% or 3%, topically applied 2 to 4 times daily or Imiquimod 5%, topically applied 3 times per week, for up to 28 days and potential prolongation for up to additional 14 days.
  Interventions: Drug: Investigator's choice
- Part D, Pritelivir (Experimental): Oral tablets, 100mg/day (400mg loading dose on day 1) for up to 28 days and potential prolongation for up to additional 14 days
  Interventions: Drug: Pritelivir
- Part E, Pritelivir (Experimental): Oral tablets, 100mg/day (400mg loading dose on day 1) for up to 28 days and potential prolongation for up to additional 14 days
  Interventions: Drug: Pritelivir
- Part F, Pritelivir (Experimental): Oral tablets, 100mg/day (400mg loading dose on day 1) for up to 28 days and potential prolongation for up to additional 14 days
  Interventions: Drug: Pritelivir

INTERVENTIONS:
Drug: Pritelivir — 100 mg oral tablets
  Arms: Part C, Pritelivir; Part D, Pritelivir; Part E, Pritelivir; Part F, Pritelivir
Drug: Investigator's choice — Foscarnet iv, 40 mg/kg BW tid or 60mg/kg bid or Cidofovir iv, 5 mg/kg BW given once weekly or Cidofovir 1% or 3%, topically applied 2 to 4 times daily or Imiquimod 5%, Solution for iv infusion or topical application
  Other Names: Foscarnet or Cidofovir or Imiquimod
  Arms: Part C,

SUMMARY:
Randomized, open-label, multi-center, comparative trial to assess the efficacy and safety in immunocompromised subjects with acyclovir resistant or acyclovir susceptible mucocutaneous HSV infection, treated with pritelivir 100 mg once daily (following a loading dose of 400 mg as first dose to rapidly reach steady-state plasma concentration) or investigators choice, which can be either foscarnet 40 mg/kg every 8 hours or 60 mg/kg every 12 hours, or Cidofovir iv 5 mg/kg body weight given once weekly, or Cidofovir 1% or 3% topical applied 2 to 4 times daily, or Imiquimod 5% topical 3 times per week) (provided the drug is nationally approved).

DETAILED DESCRIPTION:
The trial comprises 5 Parts, Part A, B, C, D, E and F.

Part A and Part B (Phase 2) have been finalised.

* Part A is a randomized, open-label, multi-center, comparative design to assess the efficacy and safety in subjects with ACV-resistant mucocutaneous HSV infection, treated with oral pritelivir or intravenous foscarnet.
* Part B is an open-label, multi-center design to assess the efficacy and safety of pritelivir in subjects with ACV-resistant-mucocutaneous HSV and who either:

  1. present with foscarnet-resistance/intolerance, or
  2. developed foscarnet resistance/intolerance during treatment in Part A (no improvement after at least 5 days of foscarnet therapy or intolerance to foscarnet requiring cessation of foscarnet treatment).

     Parts C, D, E and F (Phase 3).
* Part C is a randomized, open-label, multi-center, comparative design to assess the efficacy and safety of oral pritelivir in subjects with acyclovir resistent (ACV-R) mucocutaneous HSV episodes. Subjects with ACV-R mucocutaneous HSV infection will be randomized 1:1 to receive either oral pritelivir or Investigator's Choice.

This trial part is designed to show superiority of pritelivir against Investigator's Choice in obtaining clinical cure, ie, number of subjects with all lesions healed within 28 days.

* Part D is an open-label, multi-center design to assess the efficacy and safety of pritelivir in subjects with ACV-R mucocutaneous HSV episodes and who in addition either:

  1. present with iv foscarnet resistance/intolerance already at Screening for inclusion, or
  2. developed foscarnet resistance/intolerance during treatment in Part C (no improvement after at least 7 days of foscarnet treatment or intolerance to foscarnet requiring cessation of foscarnet treatment). Part D has been closed in June 2022.
* Part E is an open-label, multi-center design to assess the safety and efficacy of pritelivir in subjects with acyclovir susceptible (ACV-S) mucocutaneous HSV episodes, (Part E is not being conducted in Germany).
* Part F is an open-label, multi-center design to assess the efficacy and safety of pritelivir in subjects with ACV-R mucocutaneous HSV episodes and who in addition either:

  1. present with iv foscarnet resistance/intolerance already at Screening for inclusion, or
  2. developed foscarnet resistance/intolerance during treatment in Part C (no improvement after at least 7 days of foscarnet treatment or intolerance to foscarnet requiring cessation of foscarnet treatment).
  3. cannot be enrolled into Part D anymore because enrollment into Part D has been completed.

Dosing of trial medication:

Pritelivir oral tablet as single daily doses of 100 mg (following a loading dose of 400 mg as first dose)

Comparator per investigator's choice (provided the drug listed below is nationally approved):

Foscarnet intermittent infusions of 40 mg/kg every 8 hours or 60 mg/kg every 12 hours (to be adjusted in case of renal impairment) for a minimum of 1 hour duration, or Cidofovir iv infusion of 5 mg/kg body weight given once weekly, or Cidofovir 1% or 3% topical treatment, applied 2 to 4 times daily, or Imiquimod 5% topical treatment, 3 times per week.

Duration of treatment:

Until all mucocutaneous HSV lesions are healed or up to 28 days, whichever is earlier.

A prolongation up to a maximum of 42 days may be possible depending on the clinical progress.

ELIGIBILITY:
Part C inclusion criteria

1. Immunocompromised men and women of any ethnic group aged ≥16 years.

   In Canada, Germany, Belgium:

   Immunocompromised (due to conditions including but not limited to HIV infection, hematopoietic cell or solid organ transplantation, and chronic use of immunosuppressive treatment) men and women of any ethnic group aged >18 years.
2. ACV-R mucocutaneous HSV infection based on clinical failure or positive genotypic/phenotypic ACV resistance testing for current lesion. Clinical failure is defined as no improvement after oral or iv doses for at least 7 days at doses equivalent to or greater than the local agency approved high oral doses of acyclovir, valacyclovir or famciclovir.
3. Lesions accessible for visual inspection to allow assessment of lesion healing including visualization by endoscopy.
4. Willingness to use highly effective birth control.
5. Subject, and/or their legally authorized representative, (proxy consent is not permitted in Germany), must be willing and able to understand the Informed Consent Form.
6. Negative serum β-HCG (beta-human chorionic gonadotropin) test for women of child-bearing potential at Screening and a negative urine pregnancy test at Day 1.
7. Written informed consent. For subjects, who are unable to provide informed consent for whatever reason, written consent must be obtained from the legal representative, (proxy consent is not permitted in Germany).

Part D and F inclusion criteria

All inclusion criteria as for Part C, except for inclusion criterion 2, which is replaced by:

2. ACV-R and foscarnet-R mucocutaneous HSV infection based on clinical failure or positive genotypic/phenotypic resistance testing for current lesion or documented intolerance to iv foscarnet requiring cessation of foscarnet treatment or precluding foscarnet treatment.

Subjects will be able to enter Part F only after closure of enrollment in Part D.

Part E inclusion (Part E is not being conducted in Germany)

All inclusion criteria as for Part C, except for inclusion criterion 2, which is replaced by:

2. Recurrent mucocutaneous HSV infection considered ACV-S.

Part C exclusion criteria

1. Known resistance/intolerance to pritelivir or any of the excipients.
2. Previous treatment in PRIOH-1.
3. Baseline safety laboratory abnormalities.
4. History or current evidence of gastrointestinal malabsorption which, in the opinion of the Investigator, may affect the extent of absorption of pritelivir.
5. Hemodialysis for any indication and ESRD (eGFR <15 mL/min; stage 5 CKD)
6. History or current evidence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrinological, metabolic, neurological, psychiatric, or other relevant diseases.
7. Abnormalities in hematological, clinical chemical or any other laboratory variables.
8. Not able to communicate meaningfully with the Investigator and site staff.
9. Any other condition which in the opinion of the Investigator would interfere with successful completion of this clinical trial.
10. Any other important local condition.
11. Pregnant and/or breastfeeding women.
12. Having received an investigational drug in an investigational drug trial unter certain conditions.

    Part D (complete) exclusion criteria

    All exclusion criteria as for Part C, except criterion 12, which is replaced by:
13. Having received an investigational drug in an investigational trial within 7 half-lives after the last administration of this drug before initiating trial medication, except for subjects entering Part D, who have previously received foscarnet treatment in Part C of this trial.

Participation in a clinical trial without receiving other investigational drugs (eg, follow-up phase of a trial, observational study) is permitted.

Part E exclusion criteria (Part E is not being conducted in Germany)

All exclusion criteria in Part E are identical to those in Part C with the addition of:

13. Having used acyclovir, valacyclovir, or famciclovir within 3 days prior to starting pritelivir.

Part F exclusion criteria All exclusion criteria for Part D plus 13. Part D open for enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Efficacy measured by cure rate | Up to a maximum of 28 days
  Number of subjects cured (all lesions healed as assessed by the Investigator) during the treatment period of up to 28 days relative to the total number of subjects treated with trial medication in the respective treatment group.

SECONDARY OUTCOMES:
Efficacy measured by cure rate | Up to a maximum of 42 days
  Number of subjects cured (all lesions healed as assessed by the Investigator) during the treatment period of up to 42 days relative to the total number of subjects treated with trial medication in the respective treatment group.
Efficacy measured by time to lesion healing | Up to a maximum of 42 days
  Time to lesion healing, defined as complete epithelization of the mucocutaneous HSV lesion(s) within the treatment period and no appearance of new lesions, as assessed by the Investigator.
Efficacy measured by recurrence rate | At 2 months following post treatment visit, from randomization up to a maximum of 108 days
  Recurrence rate at 2 months following PoTV assessed by telephone, defined as number of subjects with a recurrence as assessed by the Investigator following 2/3 months after PoTV relative to the total number of subjects assessed for recurrence at the respective telephone call per treatment.
Efficacy measured by recurrence rate | At 3 months following post treatment visit, from randomization up to a maximum of 139 days
  Recurrence rate at 3 months following PoTV assessed by telephone, defined as number of subjects with a recurrence as assessed by the Investigator following 2/3 months after PoTV relative to the total number of subjects assessed for recurrence at the respective telephone call per treatment.
Efficacy measured by pain rate | Up to a maximum of 42 days
  Number of days with pain at lesion site relative to the total number of days with analyzable pain data through daily subject self-reporting
Efficacy measured by time to pain cessation at site of lesion | Up to a maximum of 42 days
  Starting at first dose of trial medication until pain is no longer reported by the subject (date and time)
Efficacy measured by average pain score | Up to a maximum of 42 days
  Using a single-dimensional scale assessing pain intensity through daily subject self-reporting
Efficacy measured by clinical shedding rate | From date of randomization until the date of first documented healing, assessed up to a maximum of 42 days
  Number of HSV positive swabs per subject relative to the total number of swabs collected per subject from lesion swabs taken from HSV lesion(s)
Efficacy measured by time to cessation of shedding | Up to a maximum of 42 days
  Number of days until swabs taken are negative
Efficacy measured by mean log number of HSV DNA copies | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Mean log number of HSV DNA copies on HSV DNA positive swabs from lesion(s) as detected by quantitative real-time PCR (polymerase chain reaction).
Efficacy measured by resistance to trial medication | From date of randomization until the date of post treatment visit, assessed up to a maximum of 73 days
  Resistance to trial medication for lesions not healed within the treatment period or newly appeared lesions under treatment before or at the PoTV.
Safety measured by number of subjects developing chronic kidney disease | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Chronic kidney disease
Safety measured by percentage of subjects developing chronic kidney disease | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Chronic kidney disease
Safety measured by percentage of subjects developing acute Kidney Injury | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Acute Kidney Injury (AKI) stage >1 of KDIGO (Kidney Disease: Improving Global Outcome) criteria (increase in serum creatinine by 2.0 to 2.9 times compared to baseline or urine output <0.5 mL/kg/h for >12 hours)
Safety measured by percentage of subjects developing renal impairment | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Renal impairment
Safety measured by percentage of subjects developing electrolyte abnormality | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  All abnormal values
Safety measured by percentage of subjects developing seizures | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  All seizures
Safety measured by percentage of subjects developing anemia | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Haemoglobin measurement
Safety measured by adverse events | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Incidence of Adverse Events
Safety measured by haematology | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Incidence of abnormal hematologic laboratory test results
Safety measured by lymphadenopathy | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Incidence of lymphadenopathy measured by physical examination
Safety measured by CRP (C reactive protein ) | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Incidence of CRP increase
Safety measured by cutaneous adverse events | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Incidence of cutaneous adverse events by physical examination
Safety measured by (a)PTT (partial thromboplastin time) | From date of randomization until the date of safety follow-up visit, assessed up to a maximum of 73 days
  Incidence of (a)PTT increase
Safety measured by discontinuation rate | Up to a maximum of 42 days
  Number of subjects discontinuing pritelivir or 'Inverstigator's Choice' due to AE(s) or intolerance relative to the total number of subjects treated with pritelivir or foscarnet, respectively

CONTACTS AND LOCATIONS:
Locations (70):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Metro Infectious Disease Consultants, LLC - Huntsville, Hunstville, Alabama
  - University of South Alabama, Mobile, Alabama
  - University Arizona - Department of Medicine Arizona Health Sciences Center, Tuscon, Arizona
  - City of Hope, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Division of Infectious Diseases, Sacramento, California
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Midway Immunology and Research Center (MIRC), Ft. Pierce, Florida
  - University of Florida (UF) - Division of Infectious Disease, Gainesville, Florida
  - Links Clinical Trials, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - Metro Infectious Disease Consultants - Atlanta, Decatur, Georgia
  - Metro Infectious Disease Consultants, LLC, Burr Ridge, Illinois
  - Department of Medicine J. H. Stroger Hospital of Cook County, Chicago, Illinois
  - LSU Health Baton Rouge Pulmonary Clinic, Baton Rouge, Louisiana
  - Tulane University - School of Medicine, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Lee's Summit MO United States 64086, Lee's Summit, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Kings Country Hospital Center, Brooklyn, New York
  - David H. Koch Center at Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center - Division of Infectious Diseases, Durham, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Argentina (3):
  - Hospital Rawson, Córdoba
  - Sanatorio Mayo Privado S.A., Córdoba
  - Instituto FIDES, La Plata
- Australia (2):
  - Melbourne Health - Royal Melbourne Hospital, Parkville
  - Westmead Hospital, Centre for Infectious Disease and Microbiology, Westmead
- Belgium (3):
  - AZ Sint-Jan Brugge, Bruges
  - Centre Hospitalier Universitaire Saint Pierre, Brussels
  - AZ Delta, Roeselare
- Alberta Health Services Cross Cancer Institute at the University of Alberta, Edmonton, Alberta, Canada
- France (5):
  - CHU Limoges - Centre national de reference des Herpes virus, Limoges
  - CHU de Nantes, Nantes
  - Hôpital Saint Louis - AP-HP, Paris
  - AP-HP Hopital Necker-Enfants Malades, Paris
  - AP-HP Hopital Bichat - Claude Bernard, Paris
- Georgia (2):
  - LLC Diakor, Tbilisi
  - Multiprofile Clinic Consilium Medulla LTD, Tbilisi
- Germany (3):
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Würzburg, Würzburg
- Greece (2):
  - General Hospital of Athens - Laiko, Athens
  - Regional University General Hospital of Heraklion, Heraklion
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (3):
  - Grande Ospedale Metropolitano "Bianchi Melacrino Morelli", Calabria
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Mexico (5):
  - Unidad de Investigacion CIMA SC, Chihuahua City
  - Centro de Investigacion Clinica GRAMEL S.C., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C, Durango
  - Centro de Investigacion Farmaceutica Especializado de Occidente S.C., Guadalajara
  - Arke SMO S.A. de C.V., Veracruz
- Switzerland (3):
  - Universitaetsspital Basel, Basel
  - Hopitaux universitaires de Geneve, Geneva
  - Universitaetsspital Zuerich, Zurich
- ARENSIA Exploratory Medicine LLC, Kyiv, Ukraine
- United Kingdom (3):
  - Nhs Lothian, Edinburgh
  - Research Department of Haematology, UCL Cancer Institute, London
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No